CLINICAL TRIAL: NCT04335331
Title: Prevent Diabetes Mellitus PreDM Clinical Decision Support Intervention in Community Health Centers
Brief Title: PreDM Clinical Decision Support Intervention
Acronym: PreDM_CDS
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: AllianceChicago (Other); Erie Family Health Centers (Other Government)
Responsible Party: Principal Investigator, Matthew J O'Brien, Associate Professor, Northwestern University
Other Study IDs: STU00209789
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PreDM CDS: The PreDM CDS is a passive electronic health record button that appears automatically under the Assessment/ Plan only for patients with prediabetes. When clinicians choose to click on this button, the PreDM CDS displays the last three measurements of weight, body mass index (BMI), hemoglobin A1c (HbA1c), fasting glucose, random glucose, and creatinine. This tool included order options enabling prediabetes management in a single location within the electronic health record.

SUMMARY:
Clinical practice guidelines recommend intensive lifestyle interventions and metformin to prevent or delay type 2 diabetes; yet these treatments are not routinely used among the 86 million U.S. adults with prediabetes who may benefit from them. While clinical decision support (CDS) represents an effective approach for delivering guideline-based care, the potential of this strategy to improve diabetes prevention efforts has not been definitively tested. This study developed the novel Prevent Diabetes Mellitus Clinical Decision Support (PreDM CDS) intervention and evaluated its impact on clinical outcomes.

DETAILED DESCRIPTION:
Eighty six million U.S. adults have prediabetes, and up to 75% of them will eventually develop diabetes. Landmark clinical trials have established that intensive lifestyle interventions (ILI) and metformin are safe and effective treatments to prevent or delay diabetes in adults with prediabetes and overweight/obesity. Despite being included in expert clinical guidelines, these treatments are rarely used and few studies have explored how to promote their uptake in practice. One possible approach for increasing adoption of ILI and metformin in primary care includes clinical decision support (CDS), which uses electronic systems to create tailored recommendations for evidence-based clinical care. While a large body of evidence demonstrates that CDS can improve the delivery of other recommended preventive services, this approach has not been definitively studied for ILI and metformin. The investigators plan to address this critical knowledge gap by developing and evaluating the Prevent Diabetes Mellitus Clinical Decision Support (PreDM CDS) intervention for community health center patients with prediabetes and overweight/obesity. This novel CDS engages primary care providers and clinical staff to deliver intervention components.

This study tests the potential for CDS to promote diabetes prevention and weight loss efforts in primary care. The current study objectives were to: 1) interview providers about their preferences for CDS focused on prediabetes; 2) develop a novel CDS tool, the Prediabetes CDS (PreDM CDS), promoting evidence-based care for prediabetes; and 3) conduct a pilot evaluation of the novel CDS tool using electronic health record data. Study investigators hypothesize that the proposed PreDM CDS will increase patient's adoption of ILI and metformin, producing modest weight loss and improvements in other cardiometabolic markers.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* prediabetes
* two weight measurements during the study period

Exclusion Criteria:

* The primary exclusion criterion is type 2 diabetes.
* The following additional criteria will exclude those in whom treatment is potentially harmful or outcomes assessment may be confounded: serum creatinine >1.4mg/dL in women and >1.5mg/dL in men, uncontrolled hypertension (≥180/100mmHg), prior antidiabetic medication orders, and gastric bypass surgery or pregnancy during the evaluation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who receive primary care at participating clinics and who meet the study eligibility criteria based on automated searches of the electronic health record systems will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 7424 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
A1c order | 18 Months
  Mean differences in rates of hemoglobin A1c orders between treatment arms evaluated using mixed models adjusted for clinic site, time between visits, sex, age, race/ethnicity, and baseline cardiometabolic markers.

SECONDARY OUTCOMES:
Weight | 18 Months
  Mean between group differences in weight (lbs) evaluated using mixed models adjusted for clinic site, time between visits, sex, age, race/ethnicity, and baseline cardiometabolic markers.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew O'Brien, MD, MSc, Principal Investigator — Associate Professor
Locations (1):
- Northwestern Univeristy, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No